CLINICAL TRIAL: NCT03136718
Title: The Feasibility of mHealth Technologies to Improve Hearing Aid Use and Benefit in First-time Hearing Aid Users
Brief Title: mHealth Technologies for Hearing Aid Users
Acronym: m2Hear
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 16IH003; 213341 (Other: IRAS ID); 17/EE/0117 (Other: REC)
Record Dates: First submitted 2017-04-13; First posted 2017-05-02 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Hearing Loss
Keywords: mHealth; Hearing aids; Auditory rehabilitation; Adult; Reusable Learning Object; Education; Personalised; Telehealth; Teleaudiology
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First-time hearing aid users: Individuals using hearing aids for the first-time (or if previous users, have not having worn hearing aids for more than 3 years) will have access to the mobile-enabled RLOs (mRLOs) intervention, which will be given to the participants shortly after their hearing aid is fitted.
  Interventions: Other: Mobile-enabled RLOs (mRLOs)

INTERVENTIONS:
Other: Mobile-enabled RLOs (mRLOs) — A theoretically-driven, personalised educational intervention delivered through mobile technologies based on the C2Hear (https://www.youtube.com/C2HearOnline) RLOs. The mRLO intervention will include shorter 'bite-sized' RLOs suitable for mobile technologies. This will allow a unique dynamic tailoring approach, whereby relevant mRLOs will be provided based on the user's responses to a self-evaluation filter aid, which will enable individualised, tailored learning.

SUMMARY:
This study will establish the feasibility of a theoretically-driven, personalised educational intervention delivered through mobile technologies in first-time hearing aid users. Namely, the C2Hear (https://www.youtube.com/C2HearOnline) multimedia videos, or Reusable Learning Objects (RLOs) (Ferguson et al., 2015; 2016), will be repurposed into short 'bite-sized' mobile-enabled RLOs (mRLOs).The development of the intervention will be based on a recently developed comprehensive model of health behaviour change (COM-B) (Michie et al., 2014). The intervention will be tailored to individuals' needs, and incorporate greater user interactivity and self-evaluation.

DETAILED DESCRIPTION:
Research question: Is it feasible for first-time hearing aid users to use a personalised educational intervention delivered through mobile technologies in their everyday life?

Objectives: To establish the feasibility of the intervention by evaluating delivery, accessibility, usability, acceptability, and adherence in first-time hearing aid users. To establish suitable outcome measures to evaluate the effectiveness of the intervention in a future randomised controlled trial.

Study Design: Single centre, feasibility.

Naïve first-time hearing aid users will try out the intervention away from the laboratory. Following 10-12 weeks of independent use, the investigators will assess how the participants used the intervention using a mixed-methods approach across two parallel stages:

Stage 1. The investigators will assess the feasibility of the intervention in first-time hearing aid users, who will be invited to take part in semi-structured interviews. Using the COM-B model (Michie et al., 2014) as the framework underpinning the interviews, delivery, accessibility, usability, acceptability, and adherence of the intervention will be evaluated. Transcribed audio-recordings will be analysed using thematic analysis (Braun & Clarke, 2006). A total of 15 participants is typically sufficient to achieve data saturation (the point in data collection when no new information emerges) using this qualitative methodology (Guest et al., 2006). To allow for 18% attrition (Ferguson et al., 2016), 18 patients will be. To prevent potential confounding of the interviews, participants will not be required to complete quantitative outcome measures used in stage 2.

Stage 2. The investigators will assess which outcome measures are suitable to assess the intervention in terms how well it supported users to make changes to their behaviour. First-time hearing aid users will complete outcome measures by interview. Outcomes were selected based on the World Health Organisation's International Classification of Functioning, Disability and Health (ICF) (WHO, 2001), which provides a theoretical framework upon which to measure the success of amplification using hearing aids. At least 50 participants are required to allow for sufficient between- and within-subject variability in order to calculate important change scores for each outcome measure. To allow for 18% attrition 59 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* First-time hearing aid users (or if previous users, but not having worn hearing aids for more than 3 years)
* Familiar with mobile technologies (e.g. owns a smartphone or tablet device, or uses one regularly)
* English as a first spoken language or a good understanding of English. It is important that participants can understand the content of the resources and work with the interactive elements, as well as be able to answer outcome questionnaires, to ensure valid data are collected.

Exclusion Criteria:

* Unable to complete the questionnaires without assistance due to age-related problems (e.g. cognitive decline or dementia), to ensure valid data are collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-time hearing aid users will be recruited from Nottingham Audiology Services, Nottingham University Hospitals NHS Trust, UK (secondary care). Interested patients will be invited to participate within 2 weeks of receiving their hearing aid, ideally as soon as possible. Participants will be recruited using maximum variation sampling.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Glasgow Hearing Aid Benefit Profile (GHABP: Gatehouse, 1999) - Hearing aid use | Following 10-12 weeks of independent use of the mRLO intervention
  Self-reported hearing aid use measured on a five-point scale.

SECONDARY OUTCOMES:
Hearing aid datalogging | Following 10-12 weeks of independent use of the mRLO intervention
  Hearing aid use in hours internal to the hearing aid
Glasgow Hearing Aid Benefit Profile (GHABP) | Baseline (Part I) and following 10-12 weeks of independent use of the mRLO intervention (Part II)
  Assesses hearing disability (or activity limitations) and handicap (or participation restrictions; part 1), and hearing aid use, benefit, residual disability and satisfaction (part 2). Each domain is measured on a five-point scale.
Hearing Handicap Inventory for the Elderly (HHIE: Ventry & Weinstein, 1982) | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  25-item questionnaire designed to assess the effects of hearing loss on the emotional (n = 13), and social/situational adjustment (n = 12) of older people, scored using a three-point scale (4 = yes; 2 = sometimes; 0 = no).
Social Participation Restrictions Questionnaire (SPaRQ: Heffernan et al., 2015) | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  A 19-item inventory that assesses social behaviors (9-items) and perceptions (10-items) in adults with mild-to moderate hearing loss. Each item is measured on an 11-point response scale ranging from 'Completely Disagree' at point zero to 'Completely Agree' at point ten.
Measure of Audiologic Rehabilitation Self-efficacy for Hearing Aids (MARS-HA: West & Smith, 2007) | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  Includes four subscales: basic handling, advanced handling, adjustment to hearing aids, and aided listening skills.
  Respondents indicate how confident they are that they could do the things described on an 11-point scale (0%=cannot do this, to 100%=certain I can do this).
Hearing Aid and Communication Knowledge (HACK: Ferguson et al., 2015) | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  A 20-item open-ended questionnaire that measures free recall of knowledge relevant to practical (n = 12) and psychosocial (n = 8) issues on hearing aids and communication.
Clinical Global Impression Scale - Hearing difficulties | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  A one item questionnaire to be used to identify the minimal important change score specific to each self-reported outcome measure.
Wechsler Adult Intelligence Scale (WAIS) - Digit Span (Wechsler, 1997) | Baseline and following 10-12 weeks of independent use of the mRLO intervention
  Cognitive measure of memory recall

OTHER OUTCOMES:
Adverse effects | 12 weeks
  Adverse effects arising from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Melanie A Ferguson, PhD, Principal Investigator — National Institute for Health Research Nottingham Biomedical Research Centre, UK
Locations (1):
- National Institute for Health Research Nottingham Biomedical Research Centre, Nottingham, Non-US/Non-Canadian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferguson M, Brandreth M, Brassington W, Leighton P, Wharrad H. A Randomized Controlled Trial to Evaluate the Benefits of a Multimedia Educational Program for First-Time Hearing Aid Users. Ear Hear. 2016 Mar-Apr;37(2):123-36. doi: 10.1097/AUD.0000000000000237. PMID 26565785
- [Background] Ferguson M, Brandreth M, Brassington W, Wharrad H. Information Retention and Overload in First-Time Hearing Aid Users: An Interactive Multimedia Educational Solution. Am J Audiol. 2015 Sep;24(3):329-32. doi: 10.1044/2015_AJA-14-0088. PMID 26649541
- [Background] Michie S, Atkins L, West R. The behaviour change wheel: A guide to designing interventions. 2014;London,UK:Silverback.
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006;3(2):77-101.
- [Background] Guest G, Bunce A, Johnson L. How many interviews are enough? An experiment with data saturation and variability. Field Methods. 2006;18(1):59-82.
- [Background] World Health Organization, International classification of functioning, disability and health (ICF). 2001;WHO Press:Geneva,Switzerland.
- [Background] Gatehouse S. Glasgow Hearing Aid Benefit Profile: Derivation and validation of client-centred outcome measures for hearing aid services. J Am Acad Audiol. 1999;10(2):80-103.
- [Background] Ventry IM, Weinstein BE. The hearing handicap inventory for the elderly: a new tool. Ear Hear. 1982 May-Jun;3(3):128-34. doi: 10.1097/00003446-198205000-00006. PMID 7095321
- [Background] Heffernan E, Coulson N, Henshaw H, Barry J, Ferguson MA. The development of a measure of participation in adults with hearing loss: a qualitative study of expert views. Trials. 2015;16(Suppl 1):P30.
- [Background] West RL, Smith SL. Development of a hearing aid self-efficacy questionnaire. Int J Audiol. 2007 Dec;46(12):759-71. doi: 10.1080/14992020701545898. PMID 18049965
- [Background] Wechsler, D. Wechsler Adult Intelligence Scale Third Edition. 1997;San Antonio, USA:The Psychological Corporation.
- [Derived] Maidment DW, Heyes R, Gomez R, Coulson NS, Wharrad H, Ferguson MA. Evaluating a Theoretically Informed and Cocreated Mobile Health Educational Intervention for First-Time Hearing Aid Users: Qualitative Interview Study. JMIR Mhealth Uhealth. 2020 Aug 5;8(8):e17193. doi: 10.2196/17193. PMID 32755885